CLINICAL TRIAL: NCT06737445
Title: Comparative Efficacy of Corticosteroid Injection, Extracorporeal Shock Wave Therapy, and Radiofrequency Ablation for Chronic Plantar Fasciitis: a Prospective Randomized Controlled Trial
Brief Title: Corticosteroid Injection, Extracorporeal Shock Wave Therapy, and Radiofrequency Ablation for Chronic Plantar Fasciitis:
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kars Harakani State Hospital (Other)
Responsible Party: Principal Investigator, Erdem Sahin, Medical Doctor, Kars Harakani State Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 27093
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Chronic Plantar Fasciitis
Keywords: extracorporeal shock wave therapy (ESWT); radiofrequency thermal lesioning (RTL); Chronic plantar fasciitis; corticosteroid injection (CSI)
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Radiofrequency Ablation; Cortisone; Extracorporeal Shockwave Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Radiofrequency thermal lesioning (RTL) (Active Comparator): RTL was performed as a single session using the radiofrequency ablation device (NeuroTherm JK4A; NeuroTherm Ltd, Croydon, London, England).
  Interventions: Procedure: Radiofrequency ablation alone
- Extracorporeal shock wave therapy (ESWT) (Active Comparator): Patients underwent 3 ESWT sessions applied to the plantar heel area, once a week with the same ESWT dose (15 Hz, 2000 pulse, 4.0 bar energy density) using a BTL-5000 SWT device (BTL Industries, USA).
  Interventions: Other: Extracorporeal shock wave therapy
- Corticosteroid Injection (Active Comparator): An injection of 1 ml of betamethasone 40 mg/ml and 2 ml of bupivacaine 5 mg/ml was performed.
  Interventions: Procedure: Cortisone Injection

INTERVENTIONS:
Procedure: Radiofrequency ablation alone — RTL was performed as a single session using the radiofrequency ablation device (NeuroTherm JK4A; NeuroTherm Ltd, Croydon, London, England).
  Arms: Radiofrequency thermal lesioning (RTL)
Procedure: Cortisone Injection — An injection of 1 ml of betamethasone 40 mg/ml and 2 ml of bupivacaine 5 mg/ml was performed.
  Arms: Corticosteroid Injection
Other: Extracorporeal shock wave therapy — Patients underwent 3 ESWT sessions applied to the plantar heel area, once a week with the same ESWT dose (15 Hz, 2000 pulse, 4.0 bar energy density) using a BTL-5000 SWT device (BTL Industries, USA).
  Arms: Extracorporeal shock wave therapy (ESWT)

SUMMARY:
Chronic plantar fasciitis is a prevalent condition causing persistent heel pain, often refractory to conservative treatments. This prospective randomized controlled trial aimed to compare the effectiveness of corticosteroid injection (CSI) , extracorporeal shock wave therapy (ESWT), and radiofrequency thermal lesioning (RTL) in the management of chronic plantar fasciitis.

DETAILED DESCRIPTION:
Based on the investigators' understanding of the literature there are no randomized, controlled, prospective studies comparing the therapeutic effects of CSI, ESWT and RTL for recalcitrant plantar fasciitis. In this study, the investigators investigated and compared the outcomes of three treatment techniques in participants who had exhausted conservative treatment options over the past six months.

ELIGIBILITY:
Inclusion Criteria:

* Persistant heel pain for ≥ 6 months
* No response to at least 6 weeks of conservative treatment (including at least two of the following: NSAIDs, stretching exercises, ice, heel pads, physical therapy, or night splints)
* Age ≥ 18
* BMI ≤ 35
* VAS ≥ 5 following the first step in the morning or after periods of prolonged inactivity
* Willingness to participate in the study

Exclusion Criteria:

* Previous foot or ankle surgery, major trauma
* Tumor, osteomyelitis, or complex regional pain syndrome in the affected limb
* Allergy to local anesthesia or NSAIDs
* Pregnancy or breastfeeding
* History of calcaneal fracture
* Previous cortisone injection, ESWT, or RTL for similar complaints
* BMI >35
* Age < 18
* Use of medications for neuropathic pain (Pregabalin, Gabapentin)
* Proximal nerve lesion (e.g., spinal stenosis, sciatica, tarsal tunnel syndrome)
* Regional skin or subcutaneous infections, fat pad atrophy
* History of rheumatic disease, or hematologic conditions
* History of peripheral vascular disease
* Seronegative arthropathies, heart failure, hepatic or metabolic disorders
* Pacemaker
* History of clubfoot, pes cavus, or calcaneovalgus
* Diabetic neuropathy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) scores | 1st month. 3rd month, 6th month
  Pain score (1 to 10 points)
Foot Function Index (FFI) | 1st month. 3rd month, 6th month,
  Function score (The FFI is a self-administered index consisting of 23 items divided into 3 sub-scales.)
Roles and Maudsley Score | 1st month. 3rd month, 6th month,
  The Roles and Maudsley score is an established subjective 4-point patient assessment of pain and limitations of activity (1 = excellent result with no symptoms following treatment; 2 = significant improvement from pretreatment; 3 = patient somewhat improved; 4 = poor, symptoms identical or worse than pretreatment)

CONTACTS AND LOCATIONS:
Locations (1):
- Kars Harakani State Hospital, Kars, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Erden T, Toker B, Cengiz O, Ince B, Asci S, Toprak A. Outcome of Corticosteroid Injections, Extracorporeal Shock Wave Therapy, and Radiofrequency Thermal Lesioning for Chronic Plantar Fasciitis. Foot Ankle Int. 2021 Jan;42(1):69-75. doi: 10.1177/1071100720949469. Epub 2020 Sep 3. PMID 32880199
- [Background] Liden B, Simmons M, Landsman AS. A retrospective analysis of 22 patients treated with percutaneous radiofrequency nerve ablation for prolonged moderate to severe heel pain associated with plantar fasciitis. J Foot Ankle Surg. 2009 Nov-Dec;48(6):642-7. doi: 10.1053/j.jfas.2009.05.013. Epub 2009 Jul 5. PMID 19857819
- [Background] Alshami AM, Souvlis T, Coppieters MW. A review of plantar heel pain of neural origin: differential diagnosis and management. Man Ther. 2008 May;13(2):103-11. doi: 10.1016/j.math.2007.01.014. Epub 2007 Mar 30. PMID 17400020
- [Background] Wu PT, Lee JS, Wu KC, Wu TT, Shao CJ, Liang FW, Chern TC, Su FC, Jou IM. Ultrasound-Guided Percutaneous Radiofrequency Lesioning When Treating Recalcitrant Plantar Fasciitis: Clinical Results. Ultraschall Med. 2016 Feb;37(1):56-62. doi: 10.1055/s-0034-1385466. Epub 2014 Nov 12. PMID 25389914
- [Background] Rompe JD, Furia J, Weil L, Maffulli N. Shock wave therapy for chronic plantar fasciopathy. Br Med Bull. 2007;81-82:183-208. doi: 10.1093/bmb/ldm005. Epub 2007 Apr 24. PMID 17456546